CLINICAL TRIAL: NCT05848739
Title: A Phase 1-2 Dose-escalation and Expansion Study of ST316 in Subjects With Selected Advanced Unresectable and Metastatic Solid Tumors
Brief Title: A Phase 1-2 of ST316 With Selected Advanced Unresectable and Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sapience Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ST316-101
Record Dates: First submitted 2023-03-21; First posted 2023-05-08 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Colon Cancer; Metastatic Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Bevacizumab; IFL protocol; HMPL-013; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation Phase (Experimental): The dose cohorts will be 0.5, 1, 2, 4, 8 & 12 mg/kg IV once weekly (QW)
  Interventions: Drug: ST316
- ST316 Monotherapy Colon Rectal Cancer (CRC) Expansion phase (Experimental): ST316 Monotherapy Colon Rectal Cancer (CRC) Expansion phase n=15-30
  Interventions: Drug: ST316
- ST316 & FOLFIRI/Bevacizumab Combination Colon Rectal Cancer (CRC) Expansion phase (Experimental): ST316 & FOLFIRI/Bevacizumab Combination Colon Rectal Cancer (CRC) Expansion phase Expansion phase n=15-30
  Interventions: Drug: ST316; Drug: FOLFIRI regimen & bevacizumab
- ST316 & Fruquintinib Combination CRC Expansion phase (Experimental): ST316 & Fruquintinib Combination CRC Expansion phase n=15-30
  Interventions: Drug: ST316; Drug: Fruquintinib
- ST316 & Lonsurf + Bevacizumab Combination CRC Expansion phase (Experimental): ST316 & Lonsurf & bevacizumab n=15-30
  Interventions: Drug: ST316; Drug: Lonsurf & bevacizumab

INTERVENTIONS:
Drug: ST316 — IV
Drug: FOLFIRI regimen & bevacizumab — FOLFIRI: Days 1 and 15 of each 28-day cycle:
  * irinotecan 180 mg/m2 IV over 90 minutes concurrently with
  * leucovorin 400 mg/m2 IV over 2 hours, and then
  * 5-FU bolus 400mg/m2 (up to 15 min infusion)
  * 5-FU 2400 mg/m2 IV over 46 hours
  * bevacizumab should be administered as 5mg/kg.
  Other Names: FOLFIRI
  Arms: ST316 & FOLFIRI/Bevacizumab Combination Colon Rectal Cancer (CRC) Expansion phase
Drug: Fruquintinib — 5 mg once a day for the first 21 days of a 28-day cycle
  Arms: ST316 & Fruquintinib Combination CRC Expansion phase
Drug: Lonsurf & bevacizumab — Lonsurf 35 mg/m2 twice daily on days 1-5 and days 8-12 every 28 day bevacizumab 5 mg/kg on days 1 and 15. ST316
  Arms: ST316 & Lonsurf + Bevacizumab Combination CRC Expansion phase

SUMMARY:
This is an open-label, two-part, phase 1-2 study designed to determine the safety, tolerability, PK, pharmacodynamics (PD), and proof-of-concept efficacy of ST316 administered IV in subjects with selected advanced solid tumors likely to harbor abnormalities of the WNT/β-catenin signaling pathway. The study consists of two phases: a phase 1 dose escalation/regimen exploration phase and a phase 2 expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to sign an informed consent form (ICF) and comply with the protocol and the restrictions and assessments therein.
2. Male or female ≥18 years of age.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
4. Must have a locally advanced or metastatic inoperable tumor as follows:

   1. For the dose-escalation phase: CRC, HCC, TNBC, NSCLC, OC, melanoma, CCA, and SS.
   2. For the expansion phase: CRC. Note: if additional indications and combinations are added inclusion/exclusion criteria will be updated.
5. Agrees to provide a newly obtained biopsy of an accessible lesion (if they can be biopsied based on the Investigator's assessment) prior to the start of study treatment, and to repeat biopsy once during study treatment. Tissue obtained for the biopsy must not be previously irradiated, but a new or progressing lesion in the radiation field is acceptable. Subjects without accessible lesion for biopsy must be able to provide an archival tumor tissue sample for central lab analysis.
6. In the Investigator's opinion, the subject may not derive clinical benefit from, or is ineligible for, a particular form of standard therapy on medical grounds, or the subject failed or did not tolerate one or more of other anticancer therapies:

   a. For the dose escalation phase: i. Refractory, intolerant, or refused available standard-of-care therapies. ii. Up to three previous lines of systemic anticancer therapies for metastatic disease are allowed (adjuvant or neoadjuvant setting do not count as lines of systemic therapy).

iii. Subjects with TNBC or OC with known BRCA mutations must have been previously treated with or intolerant to Food and Drug Administration (FDA) approved treatments prior to enrolling in this study (e.g., iPARP).

iv. Subjects with OC must have been treated with, refused, or were ineligible for treatment with bevacizumab to enroll.

v. Subjects with CRC tumors that are MSI-H/dMMR must have received, refused or be intolerant to a checkpoint inhibitor (CPI).

vi. Subjects with HCC must have confirmed diagnosis of inoperable hepatocellular carcinoma by histology or clinical/radiological criteria. No more than two prior lines of systemic therapy only and Child Pugh Score A or B7.

b. For the expansion phase: i. For all cohorts: Subjects with MSI-H/dMMR must have received, refused or be intolerant to a CPI.

ii. Cohort 1 ST316 monotherapy: CRC that has progressed after or on treatment with all of the following, alone or in combination, comprising a maximum of four prior lines of therapy for their advanced/metastatic disease: oxaliplatin, irinotecan, fluoropyrimidines, anti-vascular-endothelial growth factor (VEGF), anti-epidermal growth factor receptor (EGFR) targeted agents (as indicated).

iii. Cohort 2: Combination with standard of care (SOC) FOLFIRI + bevacizumab: CRC that has progressed after or on treatment with all of the following, alone or in combination, comprising a maximum of one prior line of therapy for their advanced/metastatic disease: oxaliplatin, irinotecan, fluoropyrimidines, anti-VEGF. Subjects with RAS wild-type must have been treated with an anti-EGFR targeted agent during the first line of treatment.

iv. Cohort 3: Combination with fruquintinib: CRC that has progressed after or on treatment with all of the following, alone or in combination, comprising a maximum of two prior lines of therapy for their advanced/metastatic disease: oxaliplatin, irinotecan, fluoropyrimidines or anti-VEGF Subjects with RAS wild-type must have been treated with an anti-EGFR targeted agent during the first or second line of treatment.

v. Cohort 4: Combination with Lonsurf + beva: CRC that has progressed after or on treatment with all of the following, alone or in combination, comprising a maximum of two prior lines of therapy for their advanced/metastatic disease: oxaliplatin, irinotecan, fluoropyrimidines or anti-VEGF Subjects with RAS wild-type must have been treated with an anti-EGFR targeted agent during the first or second line of treatment.

Exclusion Criteria:

1. Known hypersensitivity to ST316 or any of its excipients.
2. Known hypersensitivity to bevacizumab, 5-FU, leucovorin or irinotecan for Cohort 2, to fruquintinib for Cohort 3 and trifluridine or tipiracil for Cohort 4 in the expansion.
3. Corrected interval between Q and T wave on electrocardiogram (ECG) (QTc) > 480 msec using Fredericia's formula.
4. Symptomatic ascites or pleural effusion. A subject who is clinically stable for 4 weeks following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible.
5. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are clinically stable for at least 2 weeks prior to study entry and have no evidence of new or enlarging brain metastases. Subjects with treated brain metastases must also follow the steroid exclusion criterion (#11) listed below.
6. For expansion phase only: presence of any other active malignancy requiring systemic therapy other than the disease under study.
7. For subjects to be treated with a regimen containing bevacizumab:

   1. History of cardiac disease: congestive heart failure (CHF) ≥NYHA Class II; active coronary artery disease, myocardial infarction within 6 months prior to study entry; unevaluated new onset angina within 3 months or unstable angina (angina symptoms at rest) or cardiac arrhythmias requiring anti-arrhythmic therapy (βeta blockers or digoxin are permitted).
   2. Current uncontrolled hypertension (systolic blood pressure [BP] >150 mmHg or diastolic pressure >90 mmHg despite optimal medical management) as well as prior history of hypertensive crisis or hypertensive encephalopathy.
   3. History of arterial thrombotic or embolic events (within 6 months prior to study entry).
   4. Significant vascular disease (e.g., aortic aneurysm, aortic dissection, symptomatic peripheral vascular disease).
   5. Evidence of bleeding diathesis or clinically significant coagulopathy.
   6. Major surgical procedure (including open biopsy, significant traumatic injury, etc.) within 28 days, or anticipation of the need for major surgical procedure during the course of the study as well as minor surgical procedure (excluding placement of a vascular access device or bone marrow biopsy) within 7 days prior to study enrollment.
   7. Proteinuria at screening as demonstrated by urinalysis with proteinuria ≥2+ (subjects discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate ≤1g of protein in 24 hours to be eligible).
   8. History of abdominal fistula, gastrointestinal perforation, peptic ulcer, or intraabdominal abscess within 6 months.
   9. Ongoing serious, non-healing wound, ulcer, or bone fracture.
   10. History of reversible posterior leukoencephalopathy syndrome (RPLS).
   11. History of hypersensitivity to Chinese hamster ovary (CHO) cells or other human or humanized recombinant antibodies.

       -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
ST316 PK parameter AUCt | 3 years
  Area under the concentration-time curve over the dosing interval
ST316 Assessment DOR | 3 years
  DOR is defined for participants achieving a confirmed CR+PR as the time from the initial response of CR+PR per investigator review according to RECIST 1.1 criteria to disease progression or death of any cause, whichever occurs earlier
ST316 PK parameter Cmax | 3 years
  Maximum observed serum concentration
ST316 PK parameter t1/2 | 3 years
  half life
ST316 PK parameter AUC∞ | 3 years
  Area under the concentration-time curve over the dosing interval time from time 0 extrapolated to infinite time
ST316 PK parameter tmax. | 3 years
  The time take to reach Maximum observed serum concentration
ST316 Assessment Overall survival (OS) | 3 Years
  Overall survival (OS) is defined as time from first study treatment to death due to any cause.
ST316 Assessment Progression-free survival (PFS) | 3 Years
  Progression-free survival (PFS) is defined as time from first study treatment to a documented disease progression according to RECIST version 1.1, as determined by the investigator, or death due to any cause, whichever occurs earlier.
ST316 Assessment Objective Response Rate (ORR) | 3 Years
  ORR defined as percentage of participants with confirmed best overall response of Confirmed complete response (CR) and partial response (PR) per investigator review according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Abi Vainstein-Haras, Study Chair — CMO
Locations (11):
- United States (11):
  - University of Alabama, Birmingham, Alabama
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Sarah Cannon Research Institute - CO, Denver, Colorado
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Westchester Medical Center, Valhalla, New York
  - Duke Universtiy, Durham, North Carolina
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - Fred Hutch Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No